CLINICAL TRIAL: NCT06261177
Title: "Take-Home" Functional Electrical Stimulation for Depression: Prototype Development and Proof of Concept Clinical Trial
Brief Title: Take-home Functional Electrical Stimulation for MDD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 22-175
Record Dates: First submitted 2024-01-04; First posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: MDD
Keywords: Major Depressive Disorder; Take-home treatment; Functional Electrical Stimulation
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active FES (Experimental): 300μs long charge-balanced biphasic pulses delivered at 40 Hz, with amplitudes in the range of 5-20 mA
  Interventions: Device: Functional Electrical Stimulation (FES)
- Sham FES (Sham Comparator): Sensory stimulation (below 8 mA)
  Interventions: Device: Sham FES

INTERVENTIONS:
Device: Functional Electrical Stimulation (FES) — 45 mins per day for the duration of 4 weeks (20 sessions).
  Arms: Active FES
Device: Sham FES — Sham FES
  Arms: Sham FES

SUMMARY:
The purpose of this study is to learn whether Functional Electrical Stimulation (FES) of the facial muscles is effective in treating major depressive disorder (MDD) and to develop a model for take-home delivery.

DETAILED DESCRIPTION:
A potential novel intervention for major depressive disorder (MDD) is bilateral functional electrical stimulation (FES) of the facial muscles. The portable FES stimulator delivers electrical current to excitable tissues. Based on the preliminary work, FES can elevate mood in healthy subjects and reduce anxiety symptoms in MDD patients. The proposed study will develop a viable prototype for a "take-home" FES device and evaluate the feasibility, tolerability, and safety of FES for participants with MDD.

This is a single-site, pilot, double-blind, randomized, sham-controlled clinical trial. The trial will evaluate the feasibility, tolerability, and safety of 20 FES sessions (over 4 weeks) for MDD. Additionally, data on the preliminary therapeutic effects of 20 FES sessions for the symptoms of MDD and associated anxiety, quality of life, and sleep will be collected.

Eligible participants enrolled in this clinical trial will have a total of 28 visits. There will be 1 screening visit which will take place over the phone, 3 on-site visits (including 1 mask development visit, 1 mask delivery visit, and the last follow-up visit), and 24 Online visits (to take place over videoconference on the Zoom platform); One baseline Visit, 20 days of the FES treatment sessions, and three post-stimulation visits.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the DSM-5 criteria for unipolar MDD with a current major depressive episode (MDE) without psychotic features, with ≤ 2 failed treatment trials (non-treatment-resistant depression), as determined by a physician and validated by a MINI done by a trained research assistant
2. No change in the medication regimen or other forms of treatments (e.g., psychotherapy) for at least 4 weeks (28 days) prior to beginning the study, during the 20-session treatment period, and the 4-week post-treatment observation period. This will be established through self-report, in combination with the Antidepressant Treatment History Form (ATHF) form filled out by the participant.
3. Men and non-pregnant women aged > 18 years

Exclusion Criteria:

* 1. Paralysis of facial nerves

  2. Metallic implants or metal braces near the potential sites of electrical stimulation and any type of implanted electronic device

  3. Current fibromyalgia or currently receiving or have received repetitive transcranial magnetic stimulation (rTMS) within the last month (28 days) before screening

  4. Past or current symptoms of mania, hypomania, mixed episodes, psychotic disorders, active substance abuse, or dependence (excluding nicotine and caffeine) which will be confirmed on the MINI done by a trained research assistant

  5. Current suicidal intent or plan as demonstrated by a score of ≥ 2 on MADRS item 10

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-12-04 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the FES for MDD | 4 weeks
  The feasibility outcome defined as recruitment dropout, data completion, and protocol compliance rates.
Tolerability and safety of the FES for MDD | 4 weeks
  The tolerability and safety outcomes defined as the number and nature of adverse events and serious adverse events, to evaluate patient experience with the FES

SECONDARY OUTCOMES:
Improvement in symptoms of depression-17-item Hamilton Depression Rating Scale (HAM-D-17) | 4 weeks
  The is a semi-structured, clinician-administered interview that has been well-validated in measuring the presence and severity of depression. This scale will be administered at baseline, at the end of each treatment week, and at each follow-up visit. Decrease in total scores defined as improvement in depressive symptoms.
Improvement in symptoms of depression-16-Item Quick Inventory of Depressive Symptomatology-Self Report (QIDS-SR-16) | 4 week
  QIDS-SR-16 is a self-rated survey that has been psychometrically validated to screen for depression, using the diagnostic criteria for MDD from the DSM-IV. This self-report measure will be done at baseline, during each treatment visit, and at each follow-up visit. Decrease in total scores defined as improvement in depressive symptoms.
Improvement in symptoms of anxiety- General Anxiety Disorder (GAD-7) | 4 week
  The GAD-7 is a self-rated questionnaire for assessing generalized anxiety disorder and its severity, and will be done at baseline, during treatment visits 5, 10, 15, and 20, and at each follow-up visit. Items are ranked on a 4-point scale from 0 (not at all sure) to 3 (nearly every day), providing a total severity score from 0 to 21.
Improvement in well-being-World Health Organization-5 Well-Being Index (WHO-5) | 4 week
  The WHO-5 Well-Being Index is a self-rated scale that is designed to measure well-being over the past two weeks. This self-report measure will be done at baseline, during treatment visits 5, 10, 15, and 20, and at each follow-up visit. Participants will rate the frequency or consistency of each positive feeling on a 6-point scale from 0 (at no time) to 5 (all of the time). The sum of scores from the five items will then be multiplied by 4, representing the participant's perceived quality of life as a percentage.
Improvement in sleep quality- Pittsburgh Sleep Quality Index (PSQI) | 4 week
  The PSQI is a self-rated scale that measure sleep habits and quality. This self-report measure will be done at baseline, during treatment visits 5, 10, 15, and 20, and at each follow-up visit. This scale is broken up into seven components that assess sleep quality, latency, duration, efficiency, disturbances, medication use, and daytime dysfunction. The sum of scores from all seven components will generate a global score of 0-21, with higher scores indicating lower sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gholamali Nezhad F, Tassone VK, Demchenko I, Chen JXM, Iwasa SN, Martin J, Desai N, Naguib HE, Popovic MR, Bhat V. "Take-home" functional electrical stimulation for depression: protocol for a prototype development and proof of concept randomized controlled trial. Pilot Feasibility Stud. 2025 May 3;11(1):60. doi: 10.1186/s40814-025-01642-4. PMID 40319334